CLINICAL TRIAL: NCT04261309
Title: BACk Pain in Elders in Norway (BACE-N); A Prospective Cohort Study of Older People Visiting Primary Care With a New Episode of Back Pain
Brief Title: BACk Pain in Elders in Norway (BACE-N)
Acronym: BACE-N
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other); University of Sydney (Other); University of Rotterdam, The Netherlands (Other); University of Bergen (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Margreth Grotle, Professor, Oslo Metropolitan University
Other Study IDs: BACE
Record Dates: First submitted 2020-01-30; First posted 2020-02-07 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Back Pain
Keywords: prognosis, prognostic factors, subgroups, burden of disease,
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly with back pain in primary healthcare: Consecutive women and men 55 years of age or older who seek primary care (GP, physiotherapist or chiropractor) with a new episode of back pain (preceded by 6 months without visiting a primary care provider for similar complaints)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Since this is an observational study there will be no interference with the care given by the primary healthcare providers. However, the usual care provided by these and other healthcare utilization used by the patients during follow-up will be recorded during the follow-ups.

SUMMARY:
An international Consortium (BACk pain in Elders: BACE) was established in 2008 in order to create standardised methodology for large cohort studies and share data on the burden of back pain in older people. BACE cohort studies have been established in several countries with the primary objective to establish the clinical course and burden of back pain in elderly, to identify prognostic factors for chronic back pain and disability, and to explore usual care provided in primary care. The BACE-N is a BACE cohort study conducted in Norway, including a broad network of clinicians covering general practitioners, physiotherapists and chiropractors working in the primary healthcare. The BACE-N project will provide new knowledge on prognosis of back-related disability and pain in elderly people who seek help in the primary healthcare, the clinical course of back pain over two follow-up years, including a thorough description of healthcare utilisation and their costs, and prognostic factors that influence good or poor prognosis for these people.

DETAILED DESCRIPTION:
Back pain represent a considerable burden worldwide, and is predominantly managed in primary care. Between 2010 and 2050, the number of people aged 60 years and older will increase by 56% in developed countries, and this transition will increase the burden of chronic back disability. Most previous studies on (low) back pain have excluded people above 60 years of age, leading to a large knowledge gap regarding the prognosis of back-related disability and pain in older people and which factors influence the transition from acute to chronic stage. Further, back pain outcomes used in the few existing studies are not selected to capture the burden and characterization of back pain in older people. Therefore, the international Consortium (BACk pain in Elders: BACE) was established in 2008 in order to create standardised methodology for large cohort studies and share data on the burden of back pain in older people. BACE cohort studies have been established in several countries, also currently in Norway, with the primary objective to establish the clinical course and burden of back pain in elderly, to identify prognostic factors for chronic back pain and disability, and to explore usual care provided in primary care.

Specific aims for the BACE-N are:

1. Explore potential differences in baseline characteristics, including main domains of measurements of putative prognostic factors and outcomes, across patients who seek general practitioner, physiotherapist and chiropractor in primary care
2. Establish the 1- and 2-year clinical course (overall prognosis) and burden of back-related disability (defined as the primary outcome)
3. Establish the 1- and 2-year clinical course (overall prognosis) and burden of pain (severity, location/radiation/neurological signs, stiffness, sleep, and use of pain medication)
4. Describe usual care provided in the primary care (for the initial episode of back pain) and cost of illness due to total healthcare consumption (including secondary care such as hospitalisation and institutionalisation) and production loss during one year of follow-up
5. Assess the association between established prognostic factors in the middle-aged back pain population (comorbidity and psychosocial profile) and back-related disability at 1-and 2-years follow-up
6. Develop and validate a prognostic model for long-term back-related disability at 1- and 2-years follow-up in these people
7. Explore prognostic factors associated with persistent and/or recurrent back pain at 1- and 2 years follow-up
8. Explore prognostic factors associated with costs of illness during 1-year of follow-up
9. Establish the 1- and 2-year incidence of falls and loss of independence (Falls Efficacy Scale) and explore prognostic factors associated with falls and loss of independence during 1- and 2-year of follow-up
10. Assess the clinical course (overall prognosis) in main outcomes (disability, pain, and costs of illness) across patients who seek general practitioner, physiotherapist and chiropractor in primary care.
11. Assess gender differences in clinical course, prognostic factors and usual care in these people.

In addition to these specific aims, the BACE-N includes several methodological studies as several of the measurements from the original BACE protocol had to be translated and validated for a Norwegian context.

The study design is a prospective observational cohort study with linked methodological studies within a primary care setting, recruiting 450 patients from three main back pain health professionals; general practitioners, physiotherapists and chiropractors. The patients are followed by questionnaire at 3, 6, 12 and 24 months after inclusion. The data collected in the BACE-N adheres to the standardised methods described in the published protocol from 2011 (Scheele J, Luijsterburg PA, Ferreira ML, Maher CG, Pereira L, Peul WC, et al. Back complaints in the elders (BACE); design of cohort studies in primary care: an international consortium. BMC Musculoskelet Disord. 2011;12:193). Likewise, the statistical approach adheres to the original plan and the PROGnosis RESearch Strategy (PROGRESS), covering overall prognosis research, prognostic factor research, and prognostic model research. The methodological studies in the BACE-N are conducted in line with the COSMIN recommendations. A protocol for the BACE-N will be registered.

ELIGIBILITY:
Inclusion Criteria:

* seek primary care (GP, physiotherapist or chiropractor)
* new episode of back pain
* no visit of primary care the preceding 6 months for back pain

Exclusion Criteria:

* cognitive impairments
* difficulties speaking and writing Norwegian
* severe mobility impairments (can not attend physical examination)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from a range of general practitioners (GPs), physiotherapists (PTs), and chiropractors working in the primary care in Norway. Patients who fit the eligibility criteria and complete the consent to participate respond to a comprehensive baseline questionnaire and undergo a standardised physical examination. The questionnaire is preferably completed electronically, but a paper version is also available for patients who are not familiar with an electronic data collection.
Sampling Method: Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
the Roland Morris Disability Questionnaire | 12 months follow-up
  Scores range from 0 to 24. Higher scores indicate more severe pain and disability.
the Roland Morris Disability Questionnaire | 24 months follow-up
  Scores range from 0 to 24. Higher scores indicate more severe pain and disability.
Numerical Pain Rating Scale | 12 months follow-up
  pain severity for back and leg pain assessed on a score from 0 (no pain) to 10 (maximum pain). Back and leg pain is scored separately.
Numerical Pain Rating Scale | 24 months
  pain severity for back and leg pain assessed on a score from 0 (no pain) to 10 (maximum pain). Back and leg pain is scored separately.

SECONDARY OUTCOMES:
Overall recovery | 12 months follow-up
  Global perceived effect scale (7-point ordinal scale)
Overall recovery | 24 months follow-up
  Global perceived effect scale (7-point ordinal scale)
Costs of healthcare utilization | 12 months follow-up
  Costs summarised for type and frequency of health care, including consultations, medication, treatment, diagnostic examinations, hospitalisation/institutionalisation, and operations.
Costs of healthcare utilization | 24 months follow-up
  Costs summarised for type and frequency of health care, including consultations, medication, treatment, diagnostic examinations, hospitalisation/institutionalisation, and operations.
Number of falls during follow-up | 12 months follow-up
  number of falls, including description of cause of the fall
Number of falls during follow-up | 24 months follow-up
  number of falls, including description of cause of the fall
Insomnia | 12 months follow-up
  Bergen Insomnia Scale, 6 items assessing sleep onsent, maintenance and early morning wakening insomnia.
Insomnia | 24 months follow-up
  Bergen Insomnia Scale, 6 items assessing sleep onsent, maintenance and early morning wakening insomnia.
Symptomatic State | 12 months follow-up
  the Patient Acceptable Symptomatic State (PASS) (5-point ordinal scale)
Symptomatic State | 24 months follow-up
  the Patient Acceptable Symptomatic State (PASS) (5-point ordinal scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Tåsen og Ullevål fysioterapi, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
BACE-N is part of the international BACE consortium. We plan to share BACE-N with other BACE researchers in the Netherlands.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: from June 2021 and maximum 10 years (due to data storing policy in Norway)
Access Criteria: Only anonymous data will be shared.

REFERENCES:
- [Derived] Sannes AC, Feller D, Pripp AH, Chiarotto A, Kretz Grondahl L, Killingmo RM, Axen I, Storheim K, Grotle M, Vigdal ON. Development, internal and external validation of a prognostic model for symptom dissatisfaction among older adults with a new episode of back pain. BMJ Open. 2025 Aug 24;15(8):e102318. doi: 10.1136/bmjopen-2025-102318. PMID 40850922
- [Derived] Grondahl LK, Axen I, Stensrud S, Hoekstra T, Vigdal ON, Killingmo RM, Storheim K, Grotle M. Identifying latent subgroups in the older population seeking primary health care for a new episode of back pain - findings from the BACE-N cohort. BMC Musculoskelet Disord. 2024 Jan 13;25(1):60. doi: 10.1186/s12891-024-07163-0. PMID 38216905
- [Derived] Vigdal ON, Storheim K, Killingmo RM, Rysstad T, Pripp AH, van der Gaag W, Chiarotto A, Koes B, Grotle M. External validation and updating of prognostic prediction models for nonrecovery among older adults seeking primary care for back pain. Pain. 2023 Dec 1;164(12):2759-2768. doi: 10.1097/j.pain.0000000000002974. Epub 2023 Jul 24. PMID 37490100
- [Derived] Vigdal ON, Storheim K, Killingmo RM, Smastuen MC, Grotle M. The one-year clinical course of back-related disability and the prognostic value of comorbidity among older adults with back pain in primary care. Pain. 2023 Apr 1;164(4):e207-e216. doi: 10.1097/j.pain.0000000000002779. Epub 2022 Sep 8. PMID 36083174
- [Derived] Killingmo RM, Storheim K, van der Windt D, Zolic-Karlsson Z, Vigdal ON, Kretz L, Smastuen MC, Grotle M. Healthcare utilization and related costs among older people seeking primary care due to back pain: findings from the BACE-N cohort study. BMJ Open. 2022 Jun 20;12(6):e057778. doi: 10.1136/bmjopen-2021-057778. PMID 35725262
- [Derived] Killingmo RM, Chiarotto A, van der Windt DA, Storheim K, Bierma-Zeinstra SMA, Smastuen MC, Zolic-Karlsson Z, Vigdal ON, Koes BW, Grotle M. Modifiable prognostic factors of high costs related to healthcare utilization among older people seeking primary care due to back pain: an identification and replication study. BMC Health Serv Res. 2022 Jun 18;22(1):793. doi: 10.1186/s12913-022-08180-2. PMID 35717179
- [Derived] Vigdal ON, Storheim K, Munk Killingmo R, Smastuen MC, Grotle M. Characteristics of older adults with back pain associated with choice of first primary care provider: a cross-sectional analysis from the BACE-N cohort study. BMJ Open. 2021 Sep 17;11(9):e053229. doi: 10.1136/bmjopen-2021-053229. PMID 34535487

DOCUMENTS (2):
  • Study Protocol: Study protocol BACE-N for clinicaltrials (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT04261309/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: Merged SAP files in the BACE-N (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT04261309/Prot_SAP_007.pdf